CLINICAL TRIAL: NCT03217825
Title: Antihypertensive Effect of Different Doses of ROSTAFUROXIN in Comparison With Losartan, Assessed by Office and Ambulatory Blood Pressure Monitoring in a Hypertensive Population Selected According to a Specific Genetic Profile.
Brief Title: Antihypertensive Effect of Different Doses of Rostafuroxin in Comparison With Losartan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVT-CV-001
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — rostafuroxin; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rostafuroxin 6 micrograms capsules (Experimental): 1 capsule of ROSTAFUROXIN (6 micrograms) once a day before breakfast.
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 50 micrograms capsules (Experimental): 1 capsule of ROSTAFUROXIN (50 micrograms) once a day before breakfast.
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 500 micrograms (Experimental): 1 capsule of ROSTAFUROXIN (500 micrograms) once a day before breakfast.
  Interventions: Drug: Rostafuroxin
- Losartan 50 mg encapsulated (Active Comparator): 1 capsule containing one cpr of Losartan 50 mg once a day before breakfast.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Rostafuroxin — This is a potent, selective and safe inhibitor of this altered mechanism and has been proved to be effective in reducing blood pressure levels in Adducin mutated rat strains and in chronic Ouabain infused rat model.
  Other Names: Rosta
  Arms: Rostafuroxin 50 micrograms capsules; Rostafuroxin 500 micrograms; Rostafuroxin 6 micrograms capsules
Drug: Losartan — COZAAR (losartan potassium) is an angiotensin II receptor (type AT1) antagonist. Losartan potassium, a nonpeptide molecule, is chemically described as 2-butyl-4-chloro-1-[p-(o-1H-tetrazol-5-ylphenyl)benzyl]imidazole- 5-methanol monopotassium salt.
  Arms: Losartan 50 mg encapsulated

SUMMARY:
The principal aim of the study is to demonstrate that Rostafuroxin is able to induce a more pronounced reduction of arterial blood pressure respect to Losartan, in hypertensive patients carrying at least one of the pre-specified gene mutations. In previous studies has been demonstrated that these mutations are able to induce specific alterations inducing an increase of sodium (Na) reabsorption at renal tubular level and an increase of arterial blood pressure. Pilot studies have demonstrated that Rostafuroxin is able to reduce the impact of these alterations, and so directly reverse the increase in blood pressure.

DETAILED DESCRIPTION:
About 30% of the world adult population is affected by hypertension in industrialised countries. Elevated arterial pressure is the major cause of cardiovascular mortality and international guidelines emphasise the benefits of reducing blood pressure. The current antihypertensive strategies may reduce by 20-30% the cardiovascular risk of hypertensive patients when this efficacy is measured in clinical trials in comparison with placebo. A precise world-wide estimation of this efficacy both in term of patient burden and healthcare costs is not available; however, a recent analysis suggests that the world-wide cost of hypertension associated cardiovascular complications is around 1,000 billions dollars. Therefore, effective improvement in the diagnosis and treatment of hypertension can provide the most significant contribution to the decrease of cardiovascular mortality and reduction of the world-wide costs associated to treatment of hypertension complications.

Most of clinical trials, performed with the aim to show a reduction of the systolic blood pressure in hypertensive patients, show that reduction of systolic blood pressure is independent from the class of tested drugs as diuretics, β blockers, Ca channel blockers or inhibitors of RAS seem to have roughly the same efficacy. These findings have been used as an argument to support the notion that the antihypertensive therapy efficacy in reducing cardiovascular risk depends on the magnitude of the blood pressure fall rather than on the mechanism of action of the drug. This view contrasts with the well established notion that the secondary prevention capacity in other cardiovascular diseases differs among these classes of drugs with minor difference on the prevention of heart failure or stroke between the Ca antagonist and the other classes of drugs.

Furthermore, the recent findings on genetic of hypertension taken together with the previous data on pathophysiology of hypertension and its cardiovascular complications are consistent with the notion that a variety of heterogeneous genetic-molecular mechanisms concur to develop the rather uniform clinical picture of primary hypertension. Drugs are small molecules that produce their effects by interacting with larger molecules (proteins) whose function or reactivity may vary from one patient to another because the variations within the gene encoding them. Therefore, it is logical to postulate that the consequence of this different interaction either in term of blood pressure reduction or cardiovascular risk prevention may vary from a patient to another according to the peculiar function of the proteins involved in a given patient.

Rostafuroxin was selected during a research program aimed to synthesizing and selecting new antihypertensive compounds able to interfere with abnormalities in Na tubular reabsorption due to humoral and/or genetic mechanisms leading to essential (or genetic) hypertension. Many studies performed on the Milan hypertensive strain of rats (MHS), bearing a primary renal alteration in the ability to excrete sodium and increased blood pressure levels, showed a clear capacity of Rostafuroxin to revert these alteration, reducing systemic blood pressure.

Rostafuroxin selectively interferes with the Na-K pump correcting its functional abnormalities without interfering with other receptors involved in blood pressure regulation or hormonal homeostasis. At nanomolar concentration, rostafuroxin reduces the Na-K pump hyperactivation induced in renal cell cultures by either incubation with nanomolar ouabain concentrations or cell transfection with the 'hypertensive' variant of adducin.

Similarly, less than 1 μg/kg os of rostafuroxin is able to completely normalize both blood pressure and the increased renal Na-K pump activity in rats made hypertensive by a chronic infusion of low-dose ouabain. The antihypertensive effect of rostafuroxin is long-lasting since it is still present 24 hours after oral administration. It is not associated with changes in heart rate. Moreover, the long-term antihypertensive activity of rostafuroxin is not associated with alterations of plasma potassium, RAAS, insulin resistance, plasma lipid profile and uricemia. These findings indicate that the normalization of renal sodium handling brought about by this compound is not accompanied by the typical side effects of diuretics, such as: hypokaliemia, increased plasma levels of renin, aldosterone, triglycerides and uric acid, or insulin resistance.

Increased levels of EO and the mutated adducin are both associated with the organ complications related to hypertension, namely cardiac hypertrophy and progression toward renal insufficiency. Cardiac and renal hypertrophy is induced in rats by chronic ouabain infusion. Rostafuroxin prevents the ouabain-induced organ hypertrophy.

Rostafuroxin has shown a high safety ratio in toxicological studies and was well tolerated in previous clinical trials.

Patients with mutated adducin and increased EO plasma levels share many functional, hormonal and biochemical characteristics with MHS rats, therefore Rostafuroxin could become a first choice treatment in such patients bearing specific gene mutations and presenting high arterial blood pressure levels.

Preliminary proof of concept studies have shown ability of Rostafuroxin to reduce arterial blood pressure levels in such a patients.

ELIGIBILITY:
Inclusion Criteria:

* Signature of a written informed consent, included informed consent on genotype analysis.
* Naive hypertensive patient (new diagnosed patient, never treated before).
* Documented mild to moderate arterial hypertension: SBP comprised between 140 and 169 mmHg and DBP between 85 and 100 mmHg;
* Presence of at least one mutated genotype or combination of genotypes corresponding to the list provided in the protocol.

Exclusion Criteria:

* Known causes of secondary or severe or malignant hypertension;
* Significant renal or hepatic disease;
* Cardiac disease requiring prohibited pharmacological treatment or history of myocardial infarction within the last 6 months;
* Atrial Fibrillation or Complete Ventricle Bundle Branch Block;
* First degree AV-block exceeding 240 msec;
* Electrocardiographic evidence of left ventricular hypertrophy;
* Pregnant or nursing women or women of childbearing potential not taking anti-contraceptive medication or not utilizing a double contraceptive method;
* Concomitant therapy with medications that may affect blood pressure;
* Diabetes mellitus (fasting plasma glucose > 125 mg/dl);
* Statins treatment.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Week 9 of treatment versus baseline
  Automated sitting and standing SBP and DBP will be recorded by physician at baseline (two visits) and at week 2, 5 and 9 of treatement.
  sitting: after the patient has rested for at least 10 minutes in a quiet room. There are five consecutive sitting BP readings with a 30 to 60 seconds interval between the readings; the mean of the last three sitting BP will be used.

SECONDARY OUTCOMES:
Diastolic blood pressure | Baseline (two visits) and then at week 2, 5 and 9 of treatment
  Diastolic blood pressure measurements will be performed at the same times of the systolic blood pressure measurements, as described above
Trough-to-peak ratio on Systolic Blood Pressure | Throughout 24 hours ABPM
  Ambulatory Blood Pressure Monitoring (ABPM)will be performed throuhgout 24 hours at baseline and at week 9 of treatement. Readings will be Centralized. The Core Laboratory will be in charge for data interpretation
Number of participants with adverse events | throughout all the study period and follow-up (30 days)
  All the Adverse Events will be recorded and followed-up till their resolution. Number of Adverse Events in each group treatment will be computed, including single event frequencies and number of patients with adverse events. AEs will be collected on spontaneous reporting by patients and a number of standard safety procedure: i.e. recording of ECGs, standard blood chemistry and haematology, performed before, during and at the end of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Bianchi Giuseppe, MD, Study Director — CVie Therapeutics Limited
Locations (1):
- Cvie Therapeutics Limited, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Citterio L, Bianchi G, Scioli GA, Glorioso N, Bigazzi R, Cusi D, Staessen JA, Cavuto S, Ferrandi M, Lanzani C, Li X, Lau LF, Chiang CE, Wang TD, Wang KL, Ferrari P, Manunta P. Antihypertensive treatment guided by genetics: PEARL-HT, the randomized proof-of-concept trial comparing rostafuroxin with losartan. Pharmacogenomics J. 2021 Jun;21(3):346-358. doi: 10.1038/s41397-021-00214-y. Epub 2021 Mar 1. PMID 33649520